CLINICAL TRIAL: NCT06695819
Title: Ergonomic Evaluation of Nail Technicians With Quick Exposure Check
Brief Title: Evaluation of Nail Technicians With Quick Exposure Check
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH99
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Postural; Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study evaluated the ergonomic risks and occupational symptoms among 35 female nail technicians using the Quick Exposure Check (QEC) and the Extended Nordic Musculoskeletal Questionnaire (NMQ-E).

DETAILED DESCRIPTION:
This clinical cross-sectional study assessed 35 female nail technicians from 14 salons in four districts on the European side of Istanbul (Bahçelievler, Küçükçekmece, Beylikdüzü, and Esenyurt). Data collection included interviews, questionnaires, and ergonomic evaluations. The European Community Respiratory Health Survey and the Extended Nordic Musculoskeletal Questionnaire (NMQ-E) were used to assess symptoms, while ergonomic risks were evaluated using the Quick Exposure Check (QEC) by trained physiatrists. Following the assessments, technicians received ergonomic training on posture correction and risk prevention.

ELIGIBILITY:
Inclusion Criteria:

* Female nail technicians aged 18-40 years.
* Actively working as a nail technician for at least six months.
* Willingness to voluntarily participate in the study.

Exclusion Criteria:

* Pre-existing musculoskeletal disease diagnosis.
* Rheumatic or neurological diseases.
* Central sensitization syndromes (e.g., fibromyalgia, chronic fatigue syndrome).
* Psychiatric illnesses or mental disorders impeding communication.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The study population consisted of 35 female nail technicians aged between 18 and 40 years, working in 14 manicure salons located across four districts (Bahçelievler, Küçükçekmece, Beylikdüzü, and Esenyurt) on the European side of Istanbul. All participants were actively employed as nail technicians for at least six months and volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Quick Exposure Check (QEC) | 0 day
  Evaluates the ergonomic risk for various body regions (back, neck, wrist/hand, shoulder/arm) using the Quick Exposure Check (QEC).Higher scores indicate worse ergonomic risks.

SECONDARY OUTCOMES:
Extended Nordic Musculoskeletal Questionnaire (NMQ-E) | 0 day
  Assesses the prevalence and severity of musculoskeletal pain or discomfort in 9 body regions (e.g., neck, back, wrists).More affirmative responses indicate higher musculoskeletal symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)